CLINICAL TRIAL: NCT01742273
Title: Vitamin K1 to Slow Progression of Vascular Calcification in Hemodialysis Patients
Brief Title: Vitamin K1 to Slow Progression of Vascular Calcification in HD Patients
Acronym: VitaVasK
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Termination stopped due to low recruitment rates
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VitaVasK; 2010-021264-14 (EudraCT Number)
Record Dates: First submitted 2012-12-03; First posted 2012-12-05 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Vitamin K 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard treatment (usual care) (No Intervention): standard treatment (usual care)
- Vitamin K1 (Experimental): Vitamin K1 (phylloquinone), thrice weekly p.o. (5mg)
  Interventions: Drug: Vitamin K1

INTERVENTIONS:
Drug: Vitamin K1 — Vitamin K1 to slow vascular calcification
  Other Names: KA-Vit Tropfen (phylloquinone)
  Arms: Vitamin K1

SUMMARY:
Patients on hemodialysis (HD) exhibit an immensely increased cardiovascular mortality associated with extensive vascular calcification (VC). In the past years the development of VC was discovered to be actively regulated and as being influenced by inhibitors of calcification (e.g. matrix-Gla-protein, fetuin-A). MGP is produced by vascular smooth muscle cells and needs post-translational modification by vitamin K dependent gamma-carboxylation to be fully active. Based on the demonstration of increased PIVKA-II levels, about 97% of all HD patients exhibit insufficient carboxylation activity. We therefore aim in this randomized, controlled study to retard the progress of coronary and aortal calcification as assessed by thoracic multislice-CT by the thrice weekly administration of 5 mg vitamin K1 (phylloquinone) to about 100 HD patients over a period of 18 months.

DETAILED DESCRIPTION:
Patients on hemodialysis (HD) exhibit an immensely increased cardiovascular mortality associated with extensive vascular calcification (VC). This forms - at least partially - the reason for the excessively increased cardiovascular mortality in this population.

In the past years the development of VC was discovered to be actively regulated and as being influenced by inhibitors of calcification (e.g. matrix-Gla-protein, fetuin-A). Matrix Gla protein (MGP) is a powerful vascular wall-based inhibitor of VC. MGP is produced by vascular smooth muscle cells and needs post-translational modification by vitamin K dependent gamma-carboxylation to be fully active. The role of MGP was discovered in knock-out mice, which died from rupture of a massively calcified aorta. Functional vitamin K deficiency induced by administration of warfarin leads to the development of VC, which in turn can be inhibited by subsequent administration of vitamin K1. Warfarin inhibits the vitamin K mediated gamma-carboxylation, which leads to the production of noncarboxylated and inactive MGP (ucMGP).

Warfarin is widely used due to its inhibitory capacity on the activation of coagulation factors. Now it has been discovered that the use of vitamin K inhibitors influences vascular health: long-term use of warfarin is associated with an increased prevalence and extent of VC in the normal population and HD patients. Warfarin is also a crucial risk factor for the development of calciphylaxis, a life-threatening complication in HD patients characterised by calcified cutaneous vessels. In turn, administration of vitamin K1 was accompanied by reduced intima-media-thickness (IMT) and increased elasticity of vessels in postmenopausal women.

Based on the demonstration of increased PIVKA-II levels, about 97% of all HD patients exhibit insufficient carboxylation activity. Together with the increased VC they represent an ideal population for interventional trials in the vitamin K system. Recently we were able to demonstrate that supplementation of vitamin K1 in such patients is well tolerated, shows only very few side effects and induces a dose dependent decrease of the inactive form Dephosphorylated noncarboxylated matrix Gla protein (dpucMGP) in serum over a six weeks period. In this trial we also observed that all dialysis patients included had insufficient vitamin K serum levels, indicating no substantial influence of food intake on vitamin K deficiency. In addition, this demonstrates that all patients have insufficient vitamin K levels to facilitate adequate MGP carboxylation.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female minimum 18 years of age
* Not less than 6 months on hemodialysis
* Cardiovascular calcification percent (coronary artery volume score > 100)
* Written consent to take part in the study
* Life expectancy not less than 18 months

Exclusion Criteria:

* Known hypersensitivity against Vitamin K1
* History of thrombosis
* intake of Vitamin K
* tumor disease
* pulse >100/min (resting heart rate)
* Intake of vitamin K antagonists (e.g. Marcumar) at baseline or in the 3 months prior to baseline
* Inflammatory bowel disease
* Short-bowel syndrome
* Significant liver dysfunction
* more than one stent in one coronary artery plus one or more stents in an additional artery
* Hemoglobin < 70 g/L
* Women who are pregnant or breastfeeding
* Women without sufficient contraception
* Alcohol or drug abuse
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
* Subject unlikely to comply with protocol, e.g. uncooperative attitude, inability to return for follow-up-visits and unlikelihood of completing the study
* Participation in a parallel clinical trial or participation in another clinical trial within the previous 3 months
* Subjects who are in any state of dependency to the sponsor or the investigators
* Employees of the sponsor or the investigators
* Subjects who have been committed to an institution by legal or regulatory order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

PRIMARY OUTCOMES:
Progression of coronary artery calcification and thoracic aortic calcification | 18 months
  Progression of coronary artery calcification and thoracic aortic calcification(absolute change of the volume score at the 18-month MSCT versus the baseline MSCT)

SECONDARY OUTCOMES:
Progression of aortic valve calcification | 18 months
  Progression of aortic valve calcification (absolute change of the Agatston-Score and volume score at the 18-month MSCT versus the baseline MSCT)
Progression of mitral valve calcification | 18 months
  Progression of mitral valve calcification (absolute change of the Agatston-Score and volume score at the 18-month MSCT versus the baseline MSCT)
Mortality from any cause within 18 months after the treatment | 6 years
  Mortality from any cause within 18 months after the treatment
Major adverse cardiovascular events: myocardial infarction, stroke, acute coronary syndrome,embolism, symptom-driven revascularization, death from cardiovascular cause within 18 months after start of treatment | 6 years
  Major adverse cardiovascular events: myocardial infarction, stroke, acute coronary syndrome,embolism, symptom-driven revascularization, death from cardiovascular cause within 18 months after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen Floege, Prof. Dr., Principal Investigator — University Hospital of RWTH Aachen -Department of Medicine II, Nephrology and Clinical Immunology
Locations (13):
- Belgium (2):
  - Université catholique de Louvain - Department of Nephrology, Brussels
  - UZ Leuven, Dept. of Nephrology, Leuven
- Germany (10):
  - KfH Curatorship for Dialysis and Renal transplantation e.V., Aachen
  - University Hospital of RWTH Aachen, Department of Medicine II, Aachen
  - Clinical Center of Coburg - Department of Medical Clinic III, Nephrology, Coburg
  - MVZ DaVita Düsseldorf, Düsseldorf
  - KfH Curatorchip for Dialysis and Renal Transplantation e.V., Düsseldorf
  - University Hospital Düsseldorf - Department of Nephrology, Düsseldorf
  - MVZ Diaverum Erkelenz/ Heinsberg, Erkelenz
  - University hospital of Erlangen - Department of Medicine 4, Nephrology and Hypertension, Erlangen
  - Internistische Facharztpraxis, Abteilung Kardiologie - Nephrologie, Dialyse Geilenkirchen, Geilenkirchen
  - KfH Curatorchip for Dialysis and Renal Transplantation e.V., Stolberg
- University Hospital at Huddings, Karolinska Institute Stockholm - Department of Renal Medicine K56, Stockholm, Sweden